CLINICAL TRIAL: NCT01406132
Title: A Phase 1, Open-Label, Mass Balance Study to Evaluate the Pharmacokinetics of ASP015K After a Single Oral Dose of 14C-Labeled ASP015K in Healthy Male Subjects
Brief Title: A Study to Assess the Pharmacokinetics of ASP015K in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Clinical Trials Registry, Astellas Pharma Global Development
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 015K-CL-PK03
Record Dates: First submitted 2011-06-30; First posted 2011-08-01 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Healthy Subjects; Pharmacokinetics of ASP015K
Keywords: ASP015K; Healthy volunteers
MeSH Terms: interventions — peficitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP015K (Experimental)
  Interventions: Drug: ASP015K

INTERVENTIONS:
Drug: ASP015K — oral

SUMMARY:
The objective of this study is to evaluate pharmacokinetics, in particular the routes of excretion and extent of metabolism of ASP015K after a single oral dose of 14C-labeled ASP015K.

DETAILED DESCRIPTION:
Eligible subjects will be admitted to the clinical research unit and confined for a minimum of 8 days.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45 kg and a body mass index (BMI) between 18 and 32 kg/m2, inclusive
* The subject has been a non-smoker for at least 3 months prior to check-in
* The subject agrees to sexual abstinence, is surgically sterile (with documentation provided by a healthcare professional), or is using a medically acceptable method to prevent pregnancy during the study period
* The subject's clinical laboratory test results are within normal limits
* The subject is medically healthy, with no clinically significant medical history or abnormalities

Exclusion Criteria:

* The subject has a history of any clinically significant gastrointestinal, cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy excluding non-melanoma skin cancer
* The subject has a history of malabsorption syndrome or previous gastrointestinal surgery that could affect drug absorption or metabolism
* The subject has a recent history of irregular defecation, such as constipation or diarrhea
* The subject has a history of drug or alcohol abuse, or a positive urine screen for alcohol or drugs of abuse/illegal drugs
* The subject has had treatment with prescription drugs or complementary and alternative medicines (CAM) within 14 days prior to study drug administration, or over the counter (OTC) medication within past week
* The subject has/had a symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to clinic check in
* The subject is known positive for human immunodeficiency virus (HIV) antibody
* The subject has a positive test for hepatitis C antibody, or positive test for hepatitis B antigen (HBsAg)
* The subject has positive tuberculosis (TB) or Quantiferon Gold test
* The subject has received an experimental agent within 30 days or five half-lives, whichever is longer, prior to study drug administration
* The subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission
* The subject has had exposure to significant radiation (eg, serial x-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring) within 12 months prior to check-in
* The subject has participated in a radio-labeled-study within the last 6 months, participated in more than one other radio-labeled study within the past 12 months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2009-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic assessment through radiographic and high performance liquid chromatography (HPLC) analysis of blood, urine and feces samples | Up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Covance Clinical Research Unit (CCRU), Madison, Wisconsin, United States